CLINICAL TRIAL: NCT00455156
Title: A Multicenter, Open-label Study on the Efficacy, Cycle Control and Safety of a Contraceptive Vaginal Ring Delivering a Daily Dose of 150µg of Nestorone® and 15µg of Ethinyl Estradiol (150/15 NES/EE CVR)
Brief Title: Study of the Safety, Efficacy and Cycle Control of a Contraceptive Vaginal Ring
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Population Council (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kimberly Myer, Senior Program Director, NICHD, Premier Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCN006; CCN006 (Other: NICHD)
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Contraception
Keywords: Contraception; Vaginal Ring
MeSH Terms: interventions — ST 1435; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 150/15 NES/EE CVR (Experimental): 150 mg of Nestorone and 15 mg of ethinyl estradiol (150/15 NES/EE CVR), administered via vaginal ring, used on a 21/7 days in/out schedule for no more than one year.
  Interventions: Drug: 150 mg of Nestorone and 15 mg of ethinyl estradiol (150/15 NES/EE CVR)

INTERVENTIONS:
Drug: 150 mg of Nestorone and 15 mg of ethinyl estradiol (150/15 NES/EE CVR) — 150 mg of Nestorone and 15 mg of ethinyl estradiol (150/15 NES/EE CVR), administered via vaginal ring, used on a 21/7 days in/out schedule for no more than one year.

SUMMARY:
The purpose of this study is to evaluate the one-year data on the contraceptive efficacy and safety of the 150/15 NES/EE CVR as the basis for regulatory approvals of this CVR as a new delivery system for contraception.

DETAILED DESCRIPTION:
There continues to be a need to develop additional long-term user controlled contraceptives. Consistent with this need, contraceptive vaginal rings (CVR) delivering synthetic estrogen and progestin hormones have been developed to provide certain advantages over available methods of hormonal contraception. Scientists at the Population Council (PC) have performed preliminary 1-year studies on an investigational CVR that releases effective doses of synthetic estrogen and progestin hormones. This CVR contains ethinyl estradiol (EE), an approved, marketed hormonal product and Nestoroneâ (NES), an investigational, new chemical entity for which there are considerable clinical data from NES formulations used in transdermal systems, implants and CVRs. A potent 19-nor progesterone derivative, NES is not active orally, but is effective when administered via non-oral routes such as vaginal rings, implants, and transdermal systems. The CVR delivery system currently under investigation contains low doses of both steroids (15µg EE and 150µg NES respectively), provides a relatively steady release rate without requiring daily administration or attention to provide the desired contraceptive effect and achieve regular menstrual cycles. Because this CVR does not require daily oral intake of steroids, it avoids the daily high concentrations of steroids to which the liver is exposed when there is repetitive, once a day administration via the oral route. After insertion of the CVR into the vagina, steroids are rapidly absorbed by vaginal tissues, pass into the general circulation, achieve a steady state by day 4, and ultimately inhibit ovulation. In the beginning of the first cycle, however, there is a "burst" effect that lasts about 48 hours and is caused by accumulation of steroids on the silastic walls of the ring following storage subsequent to manufacturing. Based on in vitro studies with this CVR and preliminary pharmacokinetic studies, this effect decreases significantly in subsequent cycles. Pharmacokinetic studies to confirm this finding are ongoing. After three weeks of use, the user removes the ring for a week to induce withdrawal bleeding, and then reinserts it on a three-weeks-in/one-week-out cyclic regimen.

The progestin used in this new contraceptive system, NES, is a 19-nor progesterone derivative. It was selected for its high anti-ovulatory potency at low doses and its potential to decrease side effects usually observed with 19-nor testosterone derived progestins. In vitro studies have demonstrated that it binds selectively to progesterone receptors, and does not bind to androgen receptors. Although it binds to the glucocorticoid receptor, in vivo assays indicate no biological activity at low doses. NES also does not bind to estrogen receptors, and based on studies conducted in women using implants containing NES alone, it does not modify greatly the lipid profiles. When combined with estrogen, further data was obtained in a Phase 2, open label study comparing effects of the NES/EE CVR on estrogen-dependent liver proteins vs. those of an OC that used an androgenic progestin (LNG). Data revealed a significant increase in HDL associated with the CVR versus a decrease with the OC. In addition, data from this study demonstrated that when NES is administered vaginally with EE in the CVR, the impact on hepatic metabolism is similar to administration of EE via the oral routes with both hormonal products producing similar increases in angiotensinogen. The CVR, however, resulted in a significantly greater increase in SHBG and significantly greater decrease in protein S suggesting that due to its non-androgenic properties, NES does not counterbalance the EE effects on hepatic factors and that EE has an impact on liver proteins whether delivered vaginally or orally. Therefore, the same cautions and contraindications that apply to OCs relative to risks for thromboembolic events are likely to apply to CVRs containing EE and NES. Since there is no single marker that is known to predict such events, clinical experience and surveillance of women using new hormonal methods are required to clarify this question.

The dose selected for the CVR in the present study is based on a one-year randomized, Phase 2 clinical trial comparing three different doses, i.e. 150/15, 150/20 and 200/15µg on a 21/7 days in/out schedule. All doses showed efficacy, good bleeding control and a satisfactory safety profile, therefore the lowest effective dose, 150/15µg, was selected. Luteal activity [progesterone >10nmol/L (>3ng/ml)] occurred in 14 (12%) of 114 monitored cycles for the 50 women who comprised the group using 150/15µg dose. In a second study of 6 months duration, 150/15µg rings were used on the 21/7 vs. a 26/4-day regimen. In these two studies, users of the 150/15µg rings with the 21/7 schedules were observed for a total of 61.5 woman years. No pregnancies occurred in the 150/15µg 21/7 groups. Overall in the two studies that used this regimen, fewer than 10% of cycles measured for progesterone levels had any indication of luteal activity [progesterone >10nmol/L (>3ng/ml)], suggesting that this ring and this schedule suppresses ovulation to an effective degree. Weight was significantly correlated with luteal activity with women weighing >90kg showing increased rates of luteal activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, aged 18-<40 years who wish to use a combined hormonal contraceptive.
* Women not intending to become pregnant for 13 months.
* Intact uterus and both ovaries.
* Prior history of regular menstrual cycles of 28 ± 7 days when not using hormonal contraception; if postpartum or postabortal, history of regular menstrual cycles of 21-35 days in length and at least one cycle (2 menses) with a cycle length consistent with her past cycles.
* Sexually active (currently) and willing to discontinue current contraceptive method to participate in the study.
* In the opinion of the investigator, able to comply with the protocol, e.g. live within the study site catchment area or within a reasonable distance from the site.
* Do not meet any of the exclusion criteria.
* Signed informed consent prior to entry into the trial.

Exclusion Criteria:

* Known hypersensitivity to estrogens or progestins.
* Known hypersensitivity to silicone rubber.
* Known or suspected pregnancy.
* History of infertility of >1.0 year in woman or her male partner.
* History of vasectomy or sterility in male partner; tubal ligation (sterilization) in women
* Undiagnosed abnormal genital bleeding.
* Undiagnosed vaginal discharge or vaginal lesions or abnormalities. (Subjects diagnosed at screening with Chlamydia or gonorrhea may be included in the trial following treatment; partner treatment is also recommended. Investigators should make a determination if subjects are at high risk for reinfection, e.g. multiple sex partners, untreated partner, and whether such subjects can be included.)
* History of pelvic inflammatory disease since last pregnancy episode.
* History of toxic shock syndrome.
* Current abnormal Pap smear (women who have abnormal Paps but are ASCUS HPV negative may participate provided there is follow up for this finding per standard of care).
* Cystoceles or rectoceles or other anatomical abnormality that would preclude use of a vaginal ring.
* Women planning to undergo major surgery.
* Smoking in women who are 35 years and over or will be 35 years during the course of the trial; Women < 35 years who smoke 15 cigarettes or more must be evaluated by the PI for inclusion based on risk factors that would increase their risk for CVD, e.g. lipid levels, glucose level, BP, BMI, family history of CVD at a young age.
* Breastfeeding.
* Current or past thrombophlebitis or thromboembolic disorders.
* History of venous thrombosis or embolism in a first-degree relative <55 years of age suggesting familial defect in blood coagulation system, which in the opinion of the principal investigator, suggests use of a hormonal contraceptive could pose a significant risk.
* Cerebrovascular or cardiovascular disease.
* History of retinal vascular lesions, unexplained partial or complete loss of vision.
* Known or suspected carcinoma of the breast.
* Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia.
* Past history of any other carcinoma unless in remission for more than 5 years.
* Current or past medically diagnosed severe depression, which, in the opinion of the investigator, could be exacerbated by use of a hormonal contraceptive.
* Headaches with focal neurological symptoms.
* Severe constipation.
* History of cholestatic jaundice of pregnancy or jaundice with prior steroid use.
* Benign or malignant liver tumors; active liver disease.
* Diastolic blood pressure (BP) ³85 mm Hg and/or systolic BP ³135 mm Hg after 5-10 minutes rest.
* Known or suspected alcoholism or drug abuse.
* Abnormal serum chemistry values according to the physician's judgment.
* Participation in another clinical trial within last 30 days.
* Weight >95 kg or >209 lbs.
* Use of liver enzyme inducers on a regular basis.
* Use of monthly injectable contraceptives (e.g. cyclofem) unless suspended 2 months before initiation of treatment. Use of Depo-Proveraâ [depo-medroxyprogesterone (DMPA)] unless suspended 6 months before treatment.
* Current use of implanted hormonal contraceptives, including Mirenaâ [progestin containing intrauterine system (IUS)], Jadelleâ, Norplantâ or Implanonâ (subjects using any of these methods who request removal for reasons unrelated to the purpose of enrollment in this study may be considered for participation).
* Current use of a non-hormonal IUD. Subjects with IUDs who request removal for reasons unrelated to the purpose of enrollment in this study may be considered for participation.
* Known HIV infection.
* Women at high risk of contracting HIV, e.g. women with multiple sex partners who need to use condoms consistently, injection drug users. If women enrolled in the study do use condoms to protect against STIs, they should be instructed that this occasional use should be with non-N-9 containing condoms and they should record condom use in their diaries. Women found to have an STI at screening will be treated prior to inclusion in the study (with the exception of those infected with HIV).

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Actual)
Dates: Start 2006-12; Primary Completion 2009-01 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana L. Blithe, PH.D., Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (15):
- United States (15):
  - California Family Health Council, Los Angeles, California
  - University of Colorado - Adv. Repro. Med., Denver, Colorado
  - University of Kentucky, Lexington, Kentucky
  - Contraceptive Research and Programs, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - NYU Medical Center Family Planning Division, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - MacDonald Physicians, Inc., Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center; Division of Community Women's Health Care, Dallas, Texas
  - Jones Institute of Repro Medicine, EVMS, Norfolk, Virginia

REFERENCES:
- [Derived] Plagianos MG, Ramanadhan S, Merkatz RB, Brache V, Friedland BA, Haddad LB. Risk factors for and outcomes of ring expulsions with a 1-year contraceptive vaginal system. Am J Obstet Gynecol. 2024 May;230(5):548.e1-548.e8. doi: 10.1016/j.ajog.2024.01.020. Epub 2024 Jan 29. PMID 38295968
- [Derived] Vieira CS, Fraser IS, Plagianos MG, Burke AE, Westhoff CL, Jensen J, Brache V, Bahamondes L, Merkatz R, Sitruk-Ware R, Blithe DL. Bleeding profile associated with 1-year use of the segesterone acetate/ethinyl estradiol contraceptive vaginal system: pooled analysis from Phase 3 trials. Contraception. 2019 Dec;100(6):438-444. doi: 10.1016/j.contraception.2019.07.145. Epub 2019 Aug 6. PMID 31398307
- [Derived] Archer DF, Merkatz RB, Bahamondes L, Westhoff CL, Darney P, Apter D, Jensen JT, Brache V, Nelson AL, Banks E, Bartfai G, Portman DJ, Plagianos M, Dart C, Kumar N, Creasy GW, Sitruk-Ware R, Blithe DL. Efficacy of the 1-year (13-cycle) segesterone acetate and ethinylestradiol contraceptive vaginal system: results of two multicentre, open-label, single-arm, phase 3 trials. Lancet Glob Health. 2019 Aug;7(8):e1054-e1064. doi: 10.1016/S2214-109X(19)30265-7. Epub 2019 Jun 20. PMID 31231065
- [Derived] Huang Y, Merkatz RB, Hillier SL, Roberts K, Blithe DL, Sitruk-Ware R, Creinin MD. Effects of a One Year Reusable Contraceptive Vaginal Ring on Vaginal Microflora and the Risk of Vaginal Infection: An Open-Label Prospective Evaluation. PLoS One. 2015 Aug 12;10(8):e0134460. doi: 10.1371/journal.pone.0134460. eCollection 2015. PMID 26267119
- See also: Efficacy paper — https://pubmed.ncbi.nlm.nih.gov/31231065/
- See also: Safety paper — https://pubmed.ncbi.nlm.nih.gov/30831102/
- See also: Safety paper — https://pubmed.ncbi.nlm.nih.gov/31398307/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 150/15 NES/EE CVR
Started | 1143
Completed | 585
Not Completed | 558

BASELINE CHARACTERISTICS:
Arm/Group | 150/15 NES/EE CVR
Number analyzed (Participants) | 1143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1143
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (5.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1143
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1143

OUTCOME MEASURES:

1. Primary Outcome: Contraceptive Efficacy Using the Pearl Index for All Subjects
Description: The Pearl Index derived from using all cycles for which back up contraception is not used will be the primary efficacy endpoint. The Pearl Index is used to indicate how many women out of 100 would get pregnant using a specific birth control method over a year. It uses the formula: (Pregnancies x 12 x 100) / (Women x Months of study). The lower the Pearl Index, the more effective the contraceptive.
Time Frame: 12 Months
Population: All cycles with documented backup contraception are excluded unless the subject became pregnant in that cycle. All cycles after conception for women who became pregnant are excluded.
Measure: Number (99% Confidence Interval); unit: Number of pregnancies per 100 women mths
Units Other Than Participants: Cycles
Arm/Group | 150/15 NES/EE CVR
Number analyzed (Participants) | 1143
Number analyzed (Cycles) | 9212
Number of pregnancies per 100 women mths | 2.96 [1.93 to 4.55]

2. Primary Outcome: Changes From Baseline in Pap Smear
Description: Changes from Baseline in Pap Smear results as measured at Screening (Baseline) and at Visit 5 (Cycle 13)
Time Frame: Visit 0 and Visit 5, up to 13 months
Population: Subjects that were treated and had a pap smear performed at the respective timepoints were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | 150/15 NES/EE CVR
Number analyzed (Participants) | 1139
Participants
  Visit 0/Baseline: Normal Pap | 1060
  Visit 0/Baseline: ASCUS HPV Negative Pap | 47
  Visit 0/Baseline: Abnormal, Other Pap | 32
  Visit 5/Cycle 13: Normal Pap: number analyzed (Participants) | 744
  Visit 5/Cycle 13: Normal Pap | 629
  Visit 5/Cycle 13: ASCUS HPV Negative Pap: number analyzed (Participants) | 744
  Visit 5/Cycle 13: ASCUS HPV Negative Pap | 48
  Visit 5/Cycle 13: Abnormal, Other Pap: number analyzed (Participants) | 744
  Visit 5/Cycle 13: Abnormal, Other Pap | 67

3. Primary Outcome: Contraceptive Efficacy Using the Pearl Index for Subjects Less Than or Equal to 35 Years of Age
Description: The Pearl Index derived from using all cycles for which back up contraception is not used will be the primary efficacy endpoint and analyzed for subjects that are less than or equal to 35 years of age. The Pearl Index is used to indicate how many women out of 100 would get pregnant using a specific birth control method over a year. It uses the formula: (Pregnancies x 12 x 100) / (Women x Months of study). The lower the Pearl Index, the more effective the contraceptive.
Time Frame: 12 Months
Population: Only subjects less than or equal to 35 years of age are included in this analysis. All cycles with documented backup contraception are excluded unless the subject became pregnant in that cycle. All cycles after conception for women who became pregnant are excluded.
Measure: Number (99% Confidence Interval); unit: Number of pregnancies per 100 women mths
Units Other Than Participants: Cycles
Arm/Group | 150/15 NES/EE CVR
Number analyzed (Participants) | 1050
Number analyzed (Cycles) | 7636
Number of pregnancies per 100 women mths | 3.92 [2.60 to 5.89]

4. Secondary Outcome: Bleeding Patterns Assessed by Number of Scheduled Bleeding Days
Description: Scheduled bleeding is any bleeding or spotting that occurs during the CVR-free intervals, regardless of the duration of the regimen. The bleeding may continue into days 1-4 of the subsequent cycle. Bleeding days are assessed based on subject diaries completed during Cycles 1-13.
Time Frame: Cycles 1-13, up to 13 months
Population: subjects that completed diaries during the respective cycles are included.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 150/15 NES/EE CVR
Number analyzed (Participants) | 1143
Days
  Cycle 1: number analyzed (Participants) | 1019
  Cycle 1 | 4.3 (1.75)
  Cycle 2: number analyzed (Participants) | 983
  Cycle 2 | 4.6 (2.04)
  Cycle 3: number analyzed (Participants) | 876
  Cycle 3 | 4.5 (2.02)
  Cycle 4: number analyzed (Participants) | 851
  Cycle 4 | 4.5 (2.00)
  Cycle 5: number analyzed (Participants) | 830
  Cycle 5 | 4.4 (2.05)
  Cycle 6: number analyzed (Participants) | 737
  Cycle 6 | 4.4 (2.07)
  Cycle 7: number analyzed (Participants) | 694
  Cycle 7 | 4.4 (1.96)
  Cycle 8: number analyzed (Participants) | 667
  Cycle 8 | 4.3 (2.01)
  Cycle 9: number analyzed (Participants) | 583
  Cycle 9 | 4.4 (2.01)
  Cycle 10: number analyzed (Participants) | 518
  Cycle 10 | 4.4 (2.04)
  Cycle 11: number analyzed (Participants) | 465
  Cycle 11 | 4.5 (2.06)
  Cycle 12: number analyzed (Participants) | 425
  Cycle 12 | 4.4 (1.97)
  Cycle 13: number analyzed (Participants) | 401
  Cycle 13 | 4.1 (2.20)

5. Secondary Outcome: Bleeding Patterns Assessed by Number of Unscheduled Bleeding Days
Description: Unscheduled bleeding or spotting is any bleeding or spotting that occurs while taking active hormones with 2 exceptions: 1) Bleeding/spotting that occurs during a CVR-free interval and continues to Days 1-4 of the next active cycle is not considered unscheduled and 2) Bleeding/spotting reported during Days 1-7 of the first cycle of study CVR insertion is not considered unscheduled. Bleeding days are assessed based on subject diaries completed during Cycles 1-13.
Time Frame: Cycles 1-13, up to 13 months
Population: subjects that completed diaries during the respective cycles are included.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 150/15 NES/EE CVR
Number analyzed (Participants) | 1143
Days
  Cycle 1: number analyzed (Participants) | 1019
  Cycle 1 | 1.3 (2.91)
  Cycle 2: number analyzed (Participants) | 983
  Cycle 2 | 0.8 (2.33)
  Cycle 3: number analyzed (Participants) | 876
  Cycle 3 | 0.7 (2.05)
  Cycle 4: number analyzed (Participants) | 851
  Cycle 4 | 0.8 (2.24)
  Cycle 5: number analyzed (Participants) | 830
  Cycle 5 | 0.8 (2.05)
  Cycle 6: number analyzed (Participants) | 737
  Cycle 6 | 0.8 (2.05)
  Cycle 7: number analyzed (Participants) | 694
  Cycle 7 | 1.0 (2.42)
  Cycle 8: number analyzed (Participants) | 667
  Cycle 8 | 0.9 (2.16)
  Cycle 9: number analyzed (Participants) | 583
  Cycle 9 | 1.0 (2.20)
  Cycle 10: number analyzed (Participants) | 518
  Cycle 10 | 1.0 (2.35)
  Cycle 11: number analyzed (Participants) | 465
  Cycle 11 | 1.1 (2.59)
  Cycle 12: number analyzed (Participants) | 425
  Cycle 12 | 1.1 (2.73)
  Cycle 13: number analyzed (Participants) | 401
  Cycle 13 | 1.1 (2.53)

6. Secondary Outcome: Return to Fertility Assessed by Intended Pregnancies
Description: Women who state, during the course of the study, that they wish to discontinue to become pregnant and women who indicate, at the end of the study, that they plan to become pregnant as soon as possible will be followed for up to six months or until earlier pregnancy.
Time Frame: Up to 6 Months
Population: Women who state, during the course of the study, that they wish to discontinue to become pregnant and women who indicate, at the end of the study, that they plan to become pregnant as soon as possible will be followed for up to six months or until earlier pregnancy. Only subjects that wanted to become pregnant are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 150/15 NES/EE CVR
Number analyzed (Participants) | 18
Participants | 11

7. Secondary Outcome: Number of Participants With Return of Post-Treatment Menses Within 6 Months
Description: Women, who do not wish to become pregnant at the time of termination or end of treatment, will be followed until the time of their first post-treatment menses.
Time Frame: Up to 6 Months
Population: Women, who do not wish to become pregnant at the time of termination or end of treatment, will be followed until the time of their first post-treatment menses. Only subjects that did not want to become pregnant or use hormonal contraception are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 150/15 NES/EE CVR
Number analyzed (Participants) | 145
Participants | 138

ADVERSE EVENTS:
Time Frame: Enrollment through follow-up, up to 18 months
Arm/Group | 150/15 NES/EE CVR
All-Cause Mortality (participants affected / at risk) | 0/1143
Serious Adverse Events (participants affected / at risk) | 21/1143
Other Adverse Events (participants affected / at risk) | 1007/1143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150/15 NES/EE CVR (N=1143)
PNEUMONIA (Infections and infestations) | 2 (2)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
BIPOLAR DISORDER (Psychiatric disorders) | 1 (1)
BIPOLAR I DISORDER (Psychiatric disorders) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1)
FOOD ALLERGY (Immune system disorders) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SALIVARY GLAND ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2)
LYMPHADENITIS (Blood and lymphatic system disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
INFUSION SITE PHLEBITIS (General disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1)
UTERINE SPASM (Reproductive system and breast disorders) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)
DRUG ABUSER (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150/15 NES/EE CVR (N=1143)
NASOPHARYNGITIS (Infections and infestations) | 212 (212)
UPPER RESPIRATORY TRACK INFECTION (Infections and infestations) | 204 (204)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 142 (142)
URINARY TRACT INFECTION (Infections and infestations) | 97 (97)
INFLUENZA (Infections and infestations) | 98 (98)
SINUSITIS (Infections and infestations) | 71 (71)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 75 (75)
METTRORRHAGIA (Reproductive system and breast disorders) | 58 (58)
BREAST TENDERNESS (Respiratory, thoracic and mediastinal disorders) | 69 (69)
GENITAL PRURITUS FEMALE (Reproductive system and breast disorders) | 60 (60)
NAUSEA (Gastrointestinal disorders) | 244 (244)
VOMITING (Gastrointestinal disorders) | 117 (117)
DIARRHOEA (Gastrointestinal disorders) | 120 (120)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 92 (92)
DYSPEPSIA (Gastrointestinal disorders) | 65 (65)
STOMACH DISCOMFORT (Gastrointestinal disorders) | 59 (59)
HEADACHE (Nervous system disorders) | 496 (496)
MIGRAINE (Nervous system disorders) | 58 (58)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 114 (114)
MYALGIA (Musculoskeletal and connective tissue disorders) | 82 (82)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 56 (56)
INSOMNIA (Psychiatric disorders) | 72 (72)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 95 (95)
SEASONAL ALLERGY (Immune system disorders) | 67 (67)
Dysmenorrhoea (Reproductive system and breast disorders) | 144 (144)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No